CLINICAL TRIAL: NCT03355300
Title: A Multicenter, Open-Label, Flexible Dose Study to Assess the Long-Term Safety of Pharmaceutical Grade Synthetic Cannabidiol Oral Solution in Pediatric Patients With Treatment-Resistant Childhood Absence Seizures
Brief Title: Long-Term Safety of Pharmaceutical Grade Synthetic Cannabidiol Oral Solution in Pediatric Participants With Treatment-Resistant Childhood Absence Seizures
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insys Therapeutics filed Chapter 11 and terminated all studies.
Sponsor: Radius Pharmaceuticals, Inc. (Industry)
Collaborators: Benuvia Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INS011-17-113
Record Dates: First submitted 2017-11-09; First posted 2017-11-28 (Actual); Results first posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Childhood Absence Epilepsy
MeSH Terms: conditions — Epilepsy, Absence | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cannabidiol Oral Solution (Experimental): Cannabidiol Oral solution, dose as assigned in INS-17-103.
  Interventions: Drug: Cannabidiol Oral Solution

INTERVENTIONS:
Drug: Cannabidiol Oral Solution — An oral solution containing pharmaceutical grade cannabidiol (nonplant-based).

SUMMARY:
The primary purpose of this study is to assess the long-term safety and tolerability of Cannabidiol Oral Solution (CBD) in pediatric participants with treatment-resistant childhood absence seizures.

ELIGIBILITY:
Inclusion Criteria:

1. Completed all activities through Visit 6 (End of Study) of INS011-17-103.
2. Participant and/or parent(s)/caregiver(s) fully comprehend the informed consent form (ICF) and assent form, understand all study procedures, and can communicate satisfactorily with the investigator and study coordinator, in accordance with applicable laws, regulations, and local requirements.
3. A female participant is eligible to participate in the study if she is premenarchal, or of childbearing potential with a negative urine pregnancy test at the Screening Visit. If sexually active, she must agree to either complete abstinence from intercourse or use acceptable methods of contraception throughout the study and for 4 weeks after completion of study participation or discontinuation from investigational product.
4. A sexually active male participant or partner of enrolled participant must be willing to use acceptable methods of contraception throughout the study and for 4 weeks after completion of study participation or discontinuation from investigational product.
5. In the opinion of the investigator, the parent(s)/caregiver(s) is (are) willing and able to comply with the study procedures and visit schedules, including venipuncture, and the visit schedules.

Exclusion Criteria:

1. Participant or parent(s)/caregiver(s) have daily commitments during the study duration that would interfere with attending all study visits.
2. Experienced an anoxic episode related to study drug requiring resuscitation during their previous study.
3. Developed an adverse event thought to be related to CBD in the previous study and for whom the Investigator determines that continuing treatment with CBD would not be in the best interest of the participant.
4. Evidence of other clinically significant disease such as unstable hepatic, hematological, renal, cardiovascular, gastrointestinal, immunological, or pulmonary diseases or ongoing malignancies.
5. Compromised respiratory function or severe respiratory insufficiency.
6. Clinically significant abnormal laboratory values within the past 14 days.
7. In the opinion of the investigator, the participant is unsuitable in any other way to participate in this study.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elkashef, MD, Study Director — INSYS Therapeutics Inc
Locations (9):
- United States (9):
  - Nicklaus Children's Hospital, Miami, Florida
  - Pediatric Epilepsy and Neurology Specialists, Tampa, Florida
  - Clinical Integrative Research Center of Atlanta, Atlanta, Georgia
  - Akron Children's Hospital, Akron, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Specialty Group, Division of Child & Adolescent Neurology, Norfolk, Virginia
  - Institute for Research and Innovation | MultiCare Health System, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 11 participants who completed the INS011-17-103 study and who further received cannabidiol oral solution for this long-term safety study (INS011-17-113). Of which, 5 participants received 20 to <30 milligram/kilogram/day (mg/kg/day) and 6 participants received 30 to <40 mg/kg/day.
Groups:
- Canabidiol Oral Solution 20 to <30 mg/kg/Day: Participants who completed the INS011-17-103 further received Cannabidiol Oral Solution 20 milligrams per kilogram per day (mg/kg/day) divided twice daily (BID) for 4 weeks for a long-term safety study.
- Canabidiol Oral Solution 30 to <40 mg/kg/Day: Participants who completed the INS011-17-103 study further received Cannabidiol Oral Solution 20 mg/kg/day divided BID for 4 weeks for a long-term study.
Period: Overall Study
Arm/Group | Canabidiol Oral Solution 20 to <30 mg/kg/Day | Canabidiol Oral Solution 30 to <40 mg/kg/Day
Started | 5 | 6
Completed | 2 (One participant completed the study and 1 participant was ongoing at the time of discontinuation of the study which is neither considered completed nor discontinued.) | 4 (One participant completed the study and 3 participants were ongoing at the time of discontinuation of the study which is neither considered completed nor discontinued.)
Not Completed | 3 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Lack of Efficacy | 2 | 1
Not completed — Other reason | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled and received at least 1 dose of study drug.
Groups:
- Canabidiol Oral Solution 20 to <30 mg/kg/Day: Participants who completed the INS011-17-103 further received Cannabidiol Oral Solution 20 mg/kg/day divided BID for 4 weeks for a long-term safety study.
- Total: Total of all reporting groups
Arm/Group | Canabidiol Oral Solution 20 to <30 mg/kg/Day | Canabidiol Oral Solution 30 to <40 mg/kg/Day | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.4 (2.41) | 10.7 (3.01) | 9.6 (2.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 1 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product during the course of a clinical investigation. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product, whether or not thought to be related to the investigational product. An SAE is any untoward medical occurrence that results in death, is life-threatening, requires the participant be at a risk of death at the time of the event, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital abnormality/birth defect, or other serious event that requires medical or surgical intervention. A summary of SAEs and all other non-serious AEs, regardless of causality, is located in the Reported AEs module.
Time Frame: Baseline (Visit 6 of INS011-17-103) and Visit 10 (up to approximately 54 weeks)
Population: All participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Canabidiol Oral Solution 20 to <30 mg/kg/Day | Canabidiol Oral Solution 30 to <40 mg/kg/Day
Number analyzed (Participants) | 5 | 6
participants
  Number of participants with AEs | 5 | 4
  Number of participants with SAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline (Visit 6 of INS011-17-103) and Visit 10 (up to approximately 54 weeks)
Description: Safety population included all participants who received at least 1 dose of study medication.
Arm/Group | Canabidiol Oral Solution 20 to <30 mg/kg/Day | Canabidiol Oral Solution 30 to <40 mg/kg/Day
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 4/5 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canabidiol Oral Solution 20 to <30 mg/kg/Day (N=5) | Canabidiol Oral Solution 30 to <40 mg/kg/Day (N=6)
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Coordination abnormal (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This study was prematurely terminated by the Sponsor. Participants ongoing at the time of discontinuation of the study are neither considered completed or discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/00/NCT03355300/Prot_SAP_002.pdf